CLINICAL TRIAL: NCT06143020
Title: Effect of Erector Spinae Plane Block on Postoperative Pain in Patients With Breast Cancer Implant Reconstruction
Brief Title: Effect of ESPB on Postoperative Pain in Patients With Breast Cancer Implant Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jun Zhang, Director of the department of anaesthesiology, Shanghai cancer center, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ESPB of BCIR 2.0
Record Dates: First submitted 2021-12-06; First posted 2023-11-22 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Mammary Cancer; Erector Spinae Plane Block; Postoperative Pain
Keywords: Mammary Cancer; implant reconstruction; erector spinae plane block; Postoperative Pain
MeSH Terms: conditions — Breast Neoplasms; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector spinae plane block group (Experimental): Before surgery, an ultrasound-guided ESPB was performed. 30 mL of 0.375% ropivacaine and 0.5μ g/kg dexmedetomidine mixture was injected in the interfascial plane between rhomboideus major and erector spinae muscle.
  Ropivacaine is produced by AstraZeneca AB under the trade name of Naropin, and the specifications are 75 mg / 10 ml. Dexmedetomidine is produced by HengRui medical China and the specifications are 100μg / 1 ml。
  Interventions: Procedure: Erector spinae plane block
- Control group (No Intervention): Control groups do not receive additional analgesia.

INTERVENTIONS:
Procedure: Erector spinae plane block — In the ESPB group, the patients were placed in the lateral decubitus position. The ultrasound probe was located in longitudinal orientation at the level of the T4 spinous process and then placed 3 cm laterally from the midline to the side involved in the surgery. The ultrasound landmarks, T4 transverse process, and the overlying trapezius, rhomboideus, and erector spinae muscles, were identified. Under aseptic conditions, an 80-mm 21-gauge block needle was inserted in-plane at an angle of 30-40° in the cranial-to-caudal direction until the tip contacted the T4 transverse process.After the hydrodissection with 2-3 mL of isotonic saline solution confirmed the correct needle tip position, the intermixture was injected in the interfascial plane between rhomboideus major and erector spinae muscle. Local anesthetic spread in a fascial longitudinal pattern deep to the erector spinae muscle was visualized using ultrasound guidance.
  Other Names: Ultrasound-guided erector spinae plane block
  Arms: Erector spinae plane block group

SUMMARY:
Nowadays, the incidence of breast cancer is the first number of malignant tumors, and the primary treatment method is surgery.With the development of medical technology and concept, radical mastectomy combined breast reconstruction are becoming more and more popular.But the reconstruction caused greater trauma and more severe postoperative pain.ESPB is a new nerve block method which thought to reduce pain after thoracic and breast surgery.However, there are few studies on radical mastectomy combined breast reconstruction. So, this randomized controlled study is conducted to explore its impact on postoperative pain and thus provide more data guidance for clinical.

DETAILED DESCRIPTION:
Patients: 100 breast cancer patients who are planned radical mastectomy combined breast reconstruction Intervention: General anesthesia + erector spinae plane block Control ： General anesthesia Outcome: NRS(Numerical rating scale) of postoperative pain at the sixth hour Study:RCT

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for an radical mastectomy and implant reconstruction surgery
* Patients with American Society of Anesthesiologists (ASA) physical status I-II,
* aged 18-70 years

Exclusion Criteria:

* coagulation disorders,
* known allergy to study drugs,
* obesity (body mass index > 35 kg/m2),
* infection at the injection site,
* chronic opioid consumption, and an inability to use patient-controlled analgesia (PCA) device,
* patient refuse

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2025-08-20 (Actual); Study Completion 2025-08-25 (Actual)

PRIMARY OUTCOMES:
Post-operative acute pain score at 6 hours | 6 hours After surgery
  11-point numerical rating scale(0=no pain, 10=worst pain) at 6th hour following the surgery

SECONDARY OUTCOMES:
Postoperative quality of recovery score | 24 to 72 hours after the surgery
  The QoR-15 will be used to evaluate postoperative quality of recovery from 15 dimensions. The QoR-15 scale is a global measurement of postoperative recovery, consisting of 15 items with 10 points each, with a total score ranging from 0 (QoR very poor) to 150 (QoR very good).
Post-operative acute pain score | 1h, 12h,24, 48h, 72h after the surgery, separately.
  Pain scores at other time points except for the primary outcome. The numerical rating scale (NRS) is a line with numbers from 0 to 10 are spaced evenly across the page. And the NRS is bounded at the left-most end with "no pain" and at the right-most end with "worst pain imaginable". Pain levels below "4" are considered mild, "4-7" is moderate pain, and anything above "7" is considered severe pain. Patients are instructed to circle the number that represents the amount of pain that they are experiencing at the time of the evaluation. The movement status refers to maximum mobility of the upper arm of the surgical side. Remedial pain relief measures are initiated when the Numeric Rating Scale (NRS) score exceeds 4.
Cumulative opioid consumption after surgery | 48 hours after the surgery
  Cumulative opioid consumption after surgery
AUC of postoperative pain score | 72 hours after the surgery
  Area under the curve(AUC) of pain score 72 hours after surgery

OTHER OUTCOMES:
Number of patients with nausea and vomiting | 24 to 72 hours after the surgery
  Number of patients who experienced nausea and vomiting after surgery.
Intraoperative hemodynamic data | During the whole surgery process.
  Including mean blood pressure(mmHg), heart rate(beats/min) during the surgery.
The number of patients receiving rescue analgesia. | 24 to 72 hours after the surgery
  The number of patients receiving rescue analgesia.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhang, PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No